CLINICAL TRIAL: NCT02490761
Title: Food Intake and Preferences in Older Patients During Hospitalisation
Brief Title: Food Intake in Older Patients
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN15HN293
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Nutritional Status in Hospitalised Geriatric Patients
Keywords: Geriatrics; Nutritional Status; Hospitalisation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study cohort: Patients aged 65 years or over admitted to a geriatric ward in 2 hospitals for more than 3 days

SUMMARY:
Unintentional weight loss and undernutrition are well described problems in elderly inpatients, occurring in around 23% to 62% of hospitalised elderly in developed countries. Not only are a large number of elderly patients undernourished at admission but a substantial proportion will lose weight and become malnourished during their hospital stay, putting them at increased risk of morbidity, mortality, poor clinical outcomes and prolonged length of hospital stay. However, as it is frequently impossible to correct undernutrition prior to hospital admission, every effort should be made to prevent weight loss and correct undernutrition during hospitalization. Therefore, screening and identification of predictors of patients at risk of weight loss and undernutrition at admission, and identification of modifiable factors (e.g. eating preferences and poor food hospital intake), where intervention might be helpful, are important aspects in the management of these patients.

Before designing a food intervention study, there is a need to, firstly:

1. describe hospital food intake, eating habits and preferences in elderly inpatients during hospitalization
2. describe predictors of hospital food intake in elderly during hospitalisation
3. compare energy and protein intake in elderly inpatients during hospitalisation with the United Kingdom Dietary Reference Values (DRVs)

This study is a hospital based observational study. Eligible participants will be 125 patients (aged ≥ 65 years old) admitted to the geriatric wards of 2 hospitals in the West of Scotland. Eligible participants will be seen 96 hours after admission in order to explain the study process and to obtain written consent. The researcher will record basic body size measurements and will ask the patient questions about living conditions, feelings, memory, health, eating habits, opinions about the hospital food service. Nursing staff will be asked about patient's functional activity. The researcher will also take pictures of a subset of patients' main meals (breakfast, lunch and dinner) on a single day, prior to and after eating. The researcher will meet each patient three times in total. The first time 4 days after admission; a second time, during the hospital stay and, finally, around the time of discharge to repeat some measurements including weight, BMI, skinfold, mid upper arm circumference, grip strength and calf circumference.

ELIGIBILITY:
Inclusion Criteria:

* Screened for study participation within 96 hours after admission
* Duration of hospital admission expected to be more than 3 days
* Able to provide consent or consent obtainable from their legal representative

Exclusion Criteria:

- Receiving palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the geriatric wards at the South Glasgow University Hospital, Glasgow or the Royal Alexandra Hospital, Paisley.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2016-08-03 (Actual)

PRIMARY OUTCOMES:
Hospital food intake | Hospital admission to discharge - median 15-20 days
  Percentage of served hospital food portion consumed

SECONDARY OUTCOMES:
Predictor of hospital food intake in elderly patients | Hospital admission to discharge - median 15-20 days
  Risk of malnutrition as measured by Mini Nutritional Assessment Short Form (MNASF)
Predictor of hospital food intake in elderly patients | Hospital admission to discharge - median 15-20 days
  Functionality as measured by Barthel index of activities of daily living questionnaire
Predictor of hospital food intake in elderly patients | Hospital admission to discharge - median 15-20 days
  Mental status as measured by Mini Mental State Examination (MMSE)
Predictor of hospital food intake in elderly patients | Hospital admission to discharge - median 15-20 days
  Quality of Life as measured by "EQ-5D" questionnaire
Eating habits | Hospital admission to discharge - median 15-20 days
  As measured by Simplified Nutritional Appetite Questionnaire (SNAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Gerasimidis, PhD, Principal Investigator — University of Glasgow